CLINICAL TRIAL: NCT04999865
Title: Building Online Research Partnerships to Improve Sexual and Reproductive Health for Women With Cystic Fibrosis (CF)
Brief Title: Cystic Fibrosis Reproductive and Sexual Health Collaborative: Building Online Research Partnerships
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Emily Godfrey, Associate Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00006146
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis; Patient Engagement
Keywords: Cystic Fibrosis; Education; Patient engaged research; Training; Evaluation; Patient
MeSH Terms: conditions — Cystic Fibrosis; Patient Participation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 4-part educational program to build patient-engagement methodology capacity — We created four online training sessions. Our first training for patients/caregivers only (Research 101) was an exception, however, in which we produced a 25-minute asynchronous, self-directed learning seminar intended to be viewed before the subsequent interactive PCOR sessions. Of the three following synchronous interactive training sessions, two included both learner working groups (patients/caregivers and researchers/providers) together (PCOR 101 and PCOR Team Dynamics) and one session (PCOR Study Design) was for researchers/healthcare providers only.

SUMMARY:
This is a Patient-Centered Outcomes Research Institute engagement effort aimed at training researchers/providers and patients to work in research teams together online throughout the research process (including: development, design, and dissemination) to address critical gaps in their care. This is a change from the typical research done with people with CF as they are frequently isolated from other members of the CF community because of infection control guidelines that restrict in-person contact to avoid the spread of bacteria between patients.

This project has four aims:

1. build capacity for PCOR knowledge and skills applicable for longitudinal online engagement,
2. create and disseminate a best practices PCOR user guide for populations that solely engage online,
3. to create an interactive web-based version of our User Guide through a survey and three modified Delphi rounds, and
4. to create a comprehensive training manual for conducting PCOR online (step-by-step instructions), which will incorporate the aforementioned user guide.

DETAILED DESCRIPTION:
The CF Reproductive and Sexual Health Collaborative (CFReSHC) will introduce and support patient-centered outcomes research (PCOR) to the greater CF community using existing PCOR training products and adapt them so that they address key issues related to researcher-patient teams that solely engage online. We will create a best-practices user guide for online engagement by performing key-informant interviews with patient- or community-engaged teams and periodic assessments of day-to-day platform use with CFReSHC members and other PCOR teams.

This project has four aims:

1. build capacity for PCOR knowledge and skills applicable for longitudinal online engagement,
2. create and disseminate a best practices PCOR user guide for populations that solely engage online,
3. to create an interactive web-based version of our User Guide through a survey and three modified Delphi rounds, and
4. to create a comprehensive training manual for conducting PCOR online (step-by-step instructions), which will incorporate the aforementioned user guide.

ELIGIBILITY:
Inclusion Criteria:

* Any interested adult CF patients, CF caregivers, researchers or healthcare providers can be included in the online patient-engagement training program. Any interested patients/community members and researchers/providers involved in patient-centered outcomes reserach teams that engage online can be included for the online platform interviews.

Exclusion Criteria:

* Persons less than 18 years of age

Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants are members of the CF community (patients, caregivers, researchers, providers or other stakeholders) who have an interest in learning more about patient-engaged methodology.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge, confidence and satisfaction regarding patient-engagement methodology | four separate training programs over the course of a year
  we evaluated each of our training sessions by administering a survey to participants before the training and another similar survey immediately after the training. For both the pre- and post-training surveys, we asked participants to rate their agreement about PCOR knowledge, confidence about engaging in PCOR and training session satisfaction (post-training only) using a 5 option Likert scale. Participants were given a statement related to the learning objective and asked to rate how much they agreed with the statement with options ranging from strongly disagree, disagree, neutral, agree and strongly agree. At the end of each survey, we asked open-ended questions regarding what the participants liked about the training session and how we could improve. Surveys were administered online via REDCap.
Development of step-by-step training manual | March 2021-December 2021
  3)4) 12-15 CF and PCOR community stakeholders, selected through an application process, will attend monthly virtual meetings to provide feedback on the development of the PCOR training manual.

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Godfrey, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared

REFERENCES:
- [Derived] Godfrey EM, Thayer EK, Mentch L, Kazmerski TM, Brown G, Pam M, Al Achkar M. Development and evaluation of a virtual patient-centered outcomes research training program for the cystic fibrosis community. Res Involv Engagem. 2021 Dec 4;7(1):86. doi: 10.1186/s40900-021-00328-4. PMID 34863273